CLINICAL TRIAL: NCT06737146
Title: A Single-arm, Dose-escalation Phase I Clinical Study on Evaluating the Tolerability, Pharmacokinetic Characteristics, Safety and Preliminary Efficacy of MT027 in Patients with Recurrent or Progressive High-grade Glioma
Brief Title: Study of MT027 in Patients with Recurrent or Progressive High-grade Glioma
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Suzhou Maximum Bio-tech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MT027-HGG-002
Record Dates: First submitted 2024-12-04; First posted 2024-12-17 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: High-grade Glioma
Keywords: MT027; High-grade glioma
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- MT027 (Experimental)
  Interventions: Drug: MT027 cells suspension

INTERVENTIONS:
Drug: MT027 cells suspension — MT027: CRISPR/Cas9 edited B7H3-specific allogeneic CAR-T cells

SUMMARY:
The clinical protocol plans to preset three dose groups, namely 1×10⁷ cells per dose, 3×10⁷ cells per dose, and 6×10⁷ cells per dose. The injection will be administered once every three weeks, adopting a "3 + 3" dose escalation design. The dosing interval is based on the pharmacokinetic (PK), safety and preliminary efficacy data of MT027 investigator-initiated trial (IIT) previously conducted at Dushu Lake Hospital of Soochow University. Accordingly, it is recommended to maintain the dosing interval of once every three weeks, with a window period of ±7 days. According to past experience, the dosing cycle should be at least 6 cycles, with each cycle lasting 21 days. If patients still benefit after more than 6 cycles, they can continue to receive the medication until no further benefit is achieved. The number of treatment sessions is approximately 6 to 9 times. However, the specific number of treatment sessions will generally be determined by the investigator based on the patient's disease condition.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participate in this study and sign the informed consent form.
2. Be aged between 18 and 70 years old (including the critical values), with no gender limitation.
3. Subjects with high-grade glioma diagnosed pathologically (referring to grade 3 or 4 in the "WHO (2021) Classification of Tumors of the Central Nervous System"), who have progressive disease during standard treatment or have recurrence after standard treatment.
4. Enhanced MRI shows space-occupying lesions in the brain, and there is at least one measurable lesion (according to the iRANO 2010 version criteria).
5. The tumor tissue of the patient has positive expression of B7-H3. The subject voluntarily provides the most recent formalin-fixed paraffin-embedded (FFPE) tissue or pathological sections (at least 8 consecutive blank sections) for the detection of B7-H3 expression (immunohistochemistry, IHC).
6. Have an expected survival period of ≥ 3 months.
7. Have a Karnofsky Performance Scale (KPS) score of ≥ 70 points. -

Exclusion Criteria:

1. Patients with recurrence in the brainstem, spinal cord dissemination or extracranial metastasis; 2. The maximum diameter of a single tumor lesion is > 5 cm, or the cumulative maximum diameter of multiple lesions is > 6 cm; 3. Having received radiotherapy within 3 months before cell therapy or having received surgical treatment (except for Ommaya reservoir implantation), chemotherapy (except for lymphocyte depletion therapy), immunotherapy, molecular targeted therapy or any other anti-tumor therapy within 4 weeks before cell therapy; 4. Having participated in other drug clinical trials within 4 weeks before screening; 5. Having previously received CAR-T cell therapy; 6. Subjects with a severe allergy history to any component of the experimental drug or biological products; 7. Subjects with other primary malignancies (except for cured cervical carcinoma in situ and basal cell carcinoma of the skin); 8. Suffering from major diseases such as active systemic infection and coagulation disorders; 9. Suffering from severe insufficiency of heart, lung, liver and kidney functions; cardiac function: grade III or above according to the New York Heart Association (NYHA) criteria; liver function: grade C or above according to the Child-Pugh grading criteria; renal function: chronic kidney disease (CKD) stage 4 or above; renal insufficiency stage III or above; pulmonary function: severe respiratory failure symptoms involving other organs; 10. Subjects with severe autoimmune diseases; 11. Subjects who have previously received allogeneic tissue/solid organ transplantation; 12. Subjects who have received live vaccines within 2 weeks before the first cell therapy or who plan to receive live vaccines during the study period; 13. Subjects with active hepatitis B virus infection; or patients with hepatitis C virus infection (defined as positive HCV antibody, and those with HCV-RNA below the detection limit are allowed to enroll); or patients with human immunodeficiency virus infection (defined as positive HIV antibody); or patients with positive treponema pallidum antibody; 14. Having symptoms and signs of epilepsy or chronic intracranial hypertension that are difficult to control with drugs (for example, those using more than 500 ml of mannitol or more than 15 mg of dexamethasone or more than 80 mg of methylprednisolone or other hormones in equivalent doses per day); 15. Subjects judged by the investigator to have severe neurocognitive disorders; 16. Pregnant or lactating women; 17. Those who are considered by the investigator to be unsuitable for participating in this clinical study due to any clinical or laboratory examination abnormalities or other reasons.

-

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Adverse Events (AE) and Serious Adverse Events (SAE) | through study completion, an average of 1 year
Dose Limiting Toxicity (DLT) | 28 days
Immune effector cell-associated neurotoxicity syndrome (ICANs) | through study completion, an average of 1 year
GvHD | through study completion, an average of 1 year
CRS | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital affiliated to Tongji Medical College of Huazhong University of Science & Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No